CLINICAL TRIAL: NCT05807633
Title: Assessment on the Performance of Novosyn® in Patients Undergoing Uterus Closure in Cesarean Section. A Retrospective, Monocenter, Observational Study in Daily Practice
Brief Title: Performance of Novosyn® in Patients Undergoing Uterus Closure in Cesarean Section
Acronym: SCOTT
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: B.Braun Surgical SA (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2128
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Cesarean Section Complications; Cesarean Section; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Novosyn®: Novosyn® used in patients undergoing uterus closure in cesarean section
  Interventions: Device: Novosyn®

INTERVENTIONS:
Device: Novosyn® — Novosyn® for uterus closure in patients undergoing cesarian section

SUMMARY:
The aim of this study is to collect clinical data on the use of Novosyn® applied for the uterus closure in cesarean section. Diverse parameters have been selected to assess that the safety and effectiveness of Novosyn® is comparable to published results, where the rate of SSIs in patients undergoing uterus closure in cesarean section was 10.6%.

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* Age ≥ 18 years
* Patients undergoing one of the following gynaecologic surgeries:
* scheduled (elective) cesarean section
* cesarean section in labour
* urgent cesarean section
* Use of Novosyn® following routine clinical practice.
* Patients with available electronic health records (EHR).

Exclusion Criteria:

* Any medical or psychological disorder that, in the investigator's opinion, may interfere with the patient's ability to comply with the study procedures.
* Participation in any clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study includes women giving birth by cesarian section.
Study Population: patients undergoing uterus closure in cesarean section
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of wound complications including post-cesarean section surgical site infections (SSIs) | within the first 30 days ± 10 days following cesarean delivery.
  Incidence of wound complications including post-cesarean section surgical site infections (SSI). The documented infections include the following:
  * Organ/space surgical site infections or endometritis
  * Primary and secondary superficial incisional surgical site infections (involving the skin and subcutaneous tissue).
  * Primary and secondary deep incisional surgical site infections (involving fascial and muscle layers).
  * Severe complications of endometritis: septicemia, peritonitis, and septic thrombosis of the pelvic vessels.

SECONDARY OUTCOMES:
incidence of post-surgery complicated wound healing | within the first 30 days ± 10 days following cesarean delivery.
  Frequency of patients with complicated wound healing. Wound healing assessment includes the healing progress, skin temperature, and the presence of oedema, seroma, and/or hematoma
Incidence of reoperations/readmissions | within the first 30 days ± 10 days following cesarean delivery.
  Frequency of reoperations/readmissions
Length of Hospital Stay | up to discharge (up to 10 days after surgery)
  Mean duration of hospital stay in patients undergoing cesarean section.
Need for blood transfusion | within the first 30 days ± 10 days following cesarean delivery.
  Frequency of patients requiring blood transfusion
Incidence of Adverse device effects (ADEs) | within the first 30 days ± 10 days following cesarean delivery.
  Frequency of patients with Adverse Device Effects (ADE), defined as any adverse event related to the use of an investigational medical device, including adverse events resulting from insufficient or inadequate Instructions for Use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device and any event resulting from use error or from intentional misuse of the investigational medical device.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Bergos Sorolla, Dra., Principal Investigator — Athaia Xarxa Assistencial Universitaria de Manresa
Locations (1):
- Athaia Xarxa Assistencial Universitaria de Manresa, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No